CLINICAL TRIAL: NCT03928002
Title: 4DFlow Magnetic Resonance Imaging in Patients With Pulmonary Hypertension Associated With Congenital Heart Disease
Acronym: 4DFlowHTAPCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A00332-53
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Congenital Heart Disease; Pulmonary Arterial Hypertension
Keywords: Eisenmenger; Pulmonary arterial hypertension; Magnetic resonance imaging; 4Dflow imagery; cardiac catheterization
MeSH Terms: conditions — Heart Defects, Congenital; Pulmonary Arterial Hypertension; Eisenmenger Complex | interventions — Cardiac Catheterization

STUDY DESIGN:
Intervention Model Description: MRI 4DFlow Cardiac cathetherization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4DFlow magnetic resonance imagery (Experimental): 2D MRI, essential for diagnosis and monitoring of PAH, with an additional 8 minutes for 4D flow
  Interventions: Other: 4D Flow magnetic resonance imagery
- Cardiac catheterization (Active Comparator): cardiac catheterization procedure using the Fick method; gold standard
  Interventions: Procedure: Cardiac catheterization

INTERVENTIONS:
Other: 4D Flow magnetic resonance imagery — acquisition of anatomical, volume, right ventricular remodeling and intracardiac flow information
  Arms: 4DFlow magnetic resonance imagery
Procedure: Cardiac catheterization — pulmonary vascular resistance calculation ;
  Arms: Cardiac catheterization

SUMMARY:
Congenital heart disease is the most common congenital anomaly. The life expectancy of children with congenital heart disease has increased considerably in recent years.

Nevertheless, the evolution of these patients is marked by an increased risk of complications. Arrhythmias, heart failure, pulmonary arterial hypertension (PAH) and endocarditis may be promoted by the absence or delay of management in childhood, by residual lesions or post-operative cardiac scars and by the presence of prosthetic materials.

PAH is a common complication of congenital heart disease, especially in non-operated shunts.

PAH corresponds to an increase in pulmonary vascular resistance and mean pulmonary arterial pressure that becomes greater than 25mmHg at rest, leading to right ventricular failure and ultimately to the patient's death.

Eisenmenger's syndrome corresponds to a non-reversible pulmonary arterial hypertension with a left-right shunt initially left open, then right-left secondary to the increase in pulmonary vascular resistance, leading to cyanosis, polycythemia and multivisceral involvement. It is the most advanced form of PAH with congenital heart disease.

PAH will be suspected during echocardiographic follow-up of any patient with congenital heart disease, on the analysis of the velocity of tricuspid and/or pulmonary regurgitation flow.

Echocardiography allows the monitoring of the VD (right ventricle) function, which is the major prognostic element in PAH. Cardiac catheterization is systematically recommended and remains the gold standard to confirm the diagnosis of PAH, establish its pathophysiology and prognosis but also for the follow-up under medical treatment of these patients in tertiary centres every 6 months. Although this tool is the gold standard, rigorously performed, it remains an invasive examination often poorly experienced by patients.

4D Flow MRI is a promising imaging that allows the acquisition of anatomical, volume, right ventricular remodeling and intracardiac flow information in a single step with 2D (only 8 minutes extra), in free breathing and totally autonomous mode. Thus, at the same time as the realization of a 2D MRI, essential for the diagnosis and follow-up of PAH, with an additional 8 minutes for 4D flow, the investigators could have additional fundamental information on pulmonary cardiac output but also prognostic markers of right ventricular dysfunction turning dramatic in pulmonary vascular disease.

DETAILED DESCRIPTION:
Cardiac catheterization is systematically recommended and remains the gold standard to confirm the diagnosis of PAH, establish its pathophysiology and prognosis but also for the follow-up under medical treatment of these patients in tertiary centres every 6 months. Some centres repeat invasive hemodynamic assessment in the event of clinical aggravation before considering a change in drug management or overall management. This is the reference examination for the calculation of PVRs, an extremely rigorous methodology is required in patients with intracardiac shunt: the Fick principle must then be applied to calculate Qp. Usually, it is calculated by thermodilution but is no longer applicable in the case of intracardiac shunt, as is significant valvulopathy or massive tricuspid leakage. Qp is equal to the oxygen consumption (MVO2) divided by the difference in oxygen content (CaO2) between the pulmonary artery and the pulmonary veins (VP). Qp= MVO2/ (CaO2VP- CaO2 AP). They must be carried out with a rigorous methodology adapted on a case-by-case basis according to the anatomy and hemodynamics of the heart disease and a precise knowledge of the limits of the technique, in expert centres in PAH and congenital heart disease and must not be seen as without consequences for the patient . Although this tool is the gold standard, rigorously carried out in our reference centre, with rare accidents or potential risks, it remains an invasive examination often poorly experienced by patients .

Magnetic resonance imaging (MRI) has emerged in recent years as the reference technique for non-invasive morphological and functional evaluation of the right ventricle. It also seems relevant for the study of pulmonary arterial hemodynamics while providing prognostic values for PAH. Its regular implementation is indicated in the 2015 ESC guidelines for the diagnosis and follow-up of patients, with more particularly an injection of gadolinium for the search for myocardial fibrosis, a marker of right ventricular remodelling. Also considered are: decrease in right ventricular ejection fraction, paradoxical septal kinetics, decrease in left ventricular dimensions, compliance of the pulmonary artery (mL/mmHg) and mean flow velocity (cm/s). Carrying out this examination using conventional techniques (2D MRI) has some limitations. Extrinsic, linked to operators and observers. The quality of the examinations here depends on the quality of the acquisitions made by the radiology manipulators (sequences / section plans) as well as an adapted analysis of these cardiopathies. All of this involves a high degree of technical expertise on the part of paramedical staff, as well as expertise in congenital heart disease and cardiac imaging for medical staff. Finally, this examination has intrinsic limitations, since it does not allow the characteristics of intracardiac or vascular flows (turbulence, direction, vortex) to be explored. All this implies an examination time of about 30 minutes 4D Flow MRI is a promising imaging that allows the acquisition of anatomical, volume, right ventricular remodeling and intracardiac flow information in a single step with 2D (only 8 minutes extra), in free breathing and totally autonomous mode. It is a sequence allowing a quasi-isotopic, retrospective analysis, providing information on blood flow in the 3 planes of the space, during the cardiac cycle. It is not influenced by the quality of the medical teams and, above all, it allows an unlimited post-processing capacity. This innovative imaging method is therefore particularly suitable for the study of cardiac output such as Qp. The right ventricular volume is difficult to analyze due to the complexity of its geometry, automatic segmentation is still under development, this element seems to be a promising hemodynamic parameter since it is quantitatively calculated and seems to be correlated with the systolic function of the left ventricle and inaccessible to conventional techniques due to the particular geometry of the right ventricle. Previous studies have demonstrated the possibility of qualitative analysis of intraventricular blood flows by studying retrograde flows, vortices and their kinetic energy, which are involved in diastolic dysfunction of the right ventricle .Studies have shown that these structures can be altered in PAH dog models but also in repaired Fallot tetralogy series and Fontan type circulations .

Thus, at the same time as the realization of a 2D MRI, essential for the diagnosis and follow-up of PAH, with an additional 8 minutes for 4D flow, the investigators could have additional fundamental information on pulmonary cardiac output but also prognostic markers of right ventricular dysfunction turning dramatic in pulmonary vascular disease.

Our objective is to evaluate the contribution of 4D MRI flow imaging to the measurement of pulmonary cardiac output compared to the gold standard which is cardiac catheterization using the Fick method. But also, to compare 2D and 4D MRI flow for the evaluation of volumes, function and right ventricular remodeling, as well as the quantification of pulmonary, tricuspid and systemic flows.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 7 years old
* Patient affiliated to a social security system
* Giving their informed consent for the study (adults, parents of minors)
* Patients with PAH associated with congenital heart disease requiring cardiac catheterization and 2D MRI for the diagnosis or follow-up of PAH associated with congenital heart disease

Exclusion Criteria:

* > Patient < 7 years old

  * Pregnant woman
  * Contraindications to MRI (claustrophobia, intraocular metal foreign bodies, pacemaker, neurostimulator, cochlear implants, old heart valves)
  * Contraindication to gadolinium injection (allergy, renal failure with DFG < 30 ml/min/1.73m²)
  * Hemodynamically unstable patients
  * Refusal to participate

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Compare the evaluation of pulmonary cardiac output (Qp) by 4D Flow MRI and cardiac catheterization using the Fick method. | one year
  Define the value of 4D flow imaging in relation to cardiac catheterization in the evaluation of Qp (Cardiac Output Pulmonary)

SECONDARY OUTCOMES:
ratio of Qp/Qs flow rates by 4D Flow and cardiac catheterization Qp by 4D Flow and 2D MRI volumes and right ventricular systolic function by 4D Flow and 2D MRI | one year
  Qp/Qs by 4D Flow and cardiac catheterization Qp per 4D Flow and 2D MRI Qp/Qs by 4D Flow and 2D MRI

CONTACTS AND LOCATIONS:
Overall Officials: HASCOET SEBASTIEN, MD, Principal Investigator — Centre Chirurgical Marie Lannelongue
Locations (1):
- centre chirurgical Marie Lannelongue, Le Plessis-Robinson, France